CLINICAL TRIAL: NCT04862611
Title: Tracking Attempts of CSE, Epidural and Spinal Insertions (TRACES)
Acronym: TRACES
Status: Completed | Type: Observational
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Anthony Chau, Clinical assistant professor, University of British Columbia
Other Study IDs: TRACES
Record Dates: First submitted 2021-04-22; First posted 2021-04-28 (Actual); Last update posted 2021-10-01 (Actual); Status verified 2021-09

CONDITIONS: Neuraxial Anesthesia Charting
Keywords: neuraxial attempts; anesthetic charting; anesthetic documentation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this study is to compare observed neuraxial (Epidural, spinal, combined spinal-epidural) insertion attempts with actual documented attempts in anesthesia providers (staff, residents and fellows) at one maternal hospital. Trained research staff will document the number of neuraxial attempts before the operation, and compare this with the attempts recorded in the patient's chart. The definition of a neuraxial attempt will be determined before the study begins through a thorough literature review.

ELIGIBILITY:
Inclusion Criteria:

* Healthy parturients receiving any neuraxial procedure

Exclusion Criteria:

* Patient refusal of observation
* Provider refusal of observation

Ages: 19 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients must meet the inclusion criteria, and give verbal consent to being watched. Providers must give verbal consent to being watched
Sampling Method: Non-Probability Sample
Enrollment: 220 (Actual)
Dates: Start 2021-01-05 (Actual); Primary Completion 2021-05-05 (Actual); Study Completion 2021-05-05 (Actual)

PRIMARY OUTCOMES:
Percent accuracy of recorded neuraxial attempts | 1 day post-operatively
  Charted neuraxial attempts divided by observed neuraxial attempts

SECONDARY OUTCOMES:
Percent accuracy of recorded neuraxial redirections | 1 day post-operatively
  Charted neuraxial attempts divided by number of observed attempts and redirections
Define a neuraxial attempt | 1 month before recruitment starts
  Use thorough literature review to establish a working definition of a neuraxial attempt
Define a neuraxial redirection | 1 month before observations start
  Use thorough literature review to establish a working definition of a neuraxial redirection
Departmental consensus on a neuraxial attempt | One week after observations conclude
  Survey the department to understand how staff define a neuraxial attempt
Completeness of documentation | 1 day post-operatively
  Percentage completion of requisite charting prompts on anesthesia record

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Chau, MD, Principal Investigator — University of British Columbia
Locations (1):
- BC Women's Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared with other researchers